CLINICAL TRIAL: NCT02314871
Title: Effects of Different Types of Perioperative Analgesia on Minimal Residual Disease Development After Colon Cancer Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: Brno University Hospital (Other); Tomas Bata Hospital, Czech Republic (Other)
Responsible Party: Principal Investigator, Marian Hajduch, M.D., Ph.D., Senior Researcher, The Institute of Molecular and Translational Medicine, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAREC-1
Record Dates: First submitted 2014-12-01; First posted 2014-12-11 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Colon Cancer; Minimal Residual Disease
Keywords: perioperative analgesia; minimal residual disease; cancer recurrence; epidural; morphine; piritramide; colon; cancer; circulating cancer cells; colon cancer surgery
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm, Residual; Neoplasms | interventions — Analgesia, Epidural; Pirinitramide; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Epidural (Active Comparator): Patients will receive perioperative epidural analgesia. Drugs: bupivacaine 1.25 mg/ml and sufentanil 0.5 mcg/ml Form and frequency: continuous infusion Dosage: 4 - 14 ml/h with boluses 2 - 4 ml based on pain assessment Duration: as long as required
  Interventions: Other: Epidural analgesia
- Piritramide (Active Comparator): Patients will receive postoperative analgesia with piritramide. Drugs: piritramide 1.0 mg/ml Form and frequency: continuous infusion Dosage: 0 - 4 ml/h with boluses 2 - 4 ml based on pain assessment Duration: as long as required
  Interventions: Drug: Piritramide
- Morphine (Active Comparator): Patients will receive postoperative analgesia with morphine. Drugs: morphine 1.0 mg/ml Form and frequency: continuous infusion Dosage: 0 - 4 ml/h with boluses 2 - 4 ml based on pain assessment Duration: as long as required
  Interventions: Drug: Morphine

INTERVENTIONS:
Other: Epidural analgesia — see Arm/group description
  Other Names: Perioperative epidural analgesia
  Arms: Epidural
Drug: Piritramide — see Arm/group description
  Other Names: Postoperative piritramide analgesia
  Arms: Piritramide
Drug: Morphine — see Arm/group description
  Other Names: Postoperative morphine analgesia
  Arms: Morphine

SUMMARY:
The aim of this study is to compare the effects of three types of perioperative analgesia on the number of circulating cancer cells (representing minimal residual disease) following radical colon cancer surgery. Patients will be randomized into one of three groups. The intervention group will receive combined regional and general anesthesia during surgery and postoperative epidural analgesia. The two control groups will receive balanced general anesthesia and either morphine-based or piritramide-based postoperative analgesia. We hypothesize that epidural analgesia will be favorable to both piritramide-based and morphine-based analgesia and that piritramide-based analgesia will be favorable to morphine-based analgesia with regard to the number of circulating cancer cells and its development in the early postoperative period.

DETAILED DESCRIPTION:
Techniques of regional analgesia such as epidural analgesia may favorably influence metastasis development following cancer surgery compared to analgesia based on strong opioids such as morphine or piritramide. These beneficial effects, if present, are probably attributable to less immunosuppression of antimetastatic immune defenses.

The aim of this study is to identify techniques of perioperative analgesia with the potential to prevent metastasis development in patients undergoing open radical colon cancer surgery. In the early postoperative period, a relationship between metastasis development and the number of circulating cancer cells representing minimal residual disease has been shown. Therefore, effects of epidural, morphine-based and piritramide-based analgesia on the number of circulating cancer cells will be compared at several time points during the peroperative and early postoperative periods. The number of circulating cancer cells will be assessed in peripheral venous blood samples using real-time polymerase chain reaction. Perioperative care will be standardized and patients will be followed by clinical observation, laboratory analyses and monitoring instrumentation daily during their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open radical surgery for colon cancer (without known extension beyond colon)
* Age over 18 years
* Written informed consent

Exclusion Criteria:

* Allergy or intolerance of morphine, piritramide, marcaine, sufentanil or volatile anesthetics
* History of colon cancer resection
* Other cancer present (apart from those in complete long-term remission for minimum 6 months)
* Chronic opioid medication and/or opioid administration 7 days or less prior to surgery
* Any contraindication to thoracic epidural anesthesia/analgesia
* Systemic therapy with immunosuppressive drugs or corticoids (apart from topical and inhalational)
* Any surgery within the last 30 days (apart from minor day-case procedures) ￼￼￼￼￼ - Chronic or acute infectious disease, particularly hepatitis, AIDS, tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline number of circulating cancer cells at 3 weeks after surgery | Baseline prior to surgery, on day 2 postoperatively and three weeks after surgery
  Number of circulating cancer cells will be measured in venous blood samples. The quantitative real-time polymerase chain reaction using carcinoembryonic antigen and cytokeratine 20 as markers for circulating cancer cells will be used for minimal residual disease detection.

SECONDARY OUTCOMES:
Pain intensity assessment | 3 days postoperatively
  Self reported pain intensity. Scale: 0 = no pain, 10 = worst pain imaginable. A score 0-10 will be recorded every four hours.

CONTACTS AND LOCATIONS:
Overall Officials: Emil Berta, MD PhD, Principal Investigator — The Institute of Molecular and Translational Medicine
Locations (2):
- Czechia (2):
  - Brno University Hospital, Brno, South Moravian
  - T. Bata Regional Hospital Zlin, Zlin, South Moravian

REFERENCES:
- See also: The Institute of Molecular and Translational Medicine, Faculty of Medicine and Dentistry Palacky University Olomouc — http://imtm.cz